CLINICAL TRIAL: NCT06374277
Title: Pharmacy-led Transitions of Care Intervention to Address System-Level Barriers and Improve Medication Adherence in Socioeconomically Disadvantaged Populations
Brief Title: Pharmacy-led Transitions of Care Intervention to Improve Medication Adherence
Acronym: MedAAAction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-09339-IAA
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Diabetes; Hypertension; High Cholesterol/Hyperlipidemia; Coronary Artery Disease; Congestive Heart Failure; Chronic Lung Disease; Chronic Kidney Diseases; Arrythmia; Stroke; Depression; Anxiety; Pulmonary Embolism; Heart Attack
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hypercholesterolemia; Hyperlipidemias; Coronary Artery Disease; Heart Failure; Renal Insufficiency, Chronic; Arrhythmias, Cardiac; Stroke; Depression; Anxiety Disorders; Pulmonary Embolism; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Eligible patients who sign consent forms and complete baseline surveys will be randomized to the Med AAAction intervention group or the usual care in a 1:1 ratio, stratified by health system. The participants will be enrolled before hospital discharge. The Med AAAction intervention will include the following components: 1) medications with zero copay, 2) bedside delivery and subsequent home delivery of medications, and 3) care coordination provided by certified pharmacy technicians/health coaches to assist with medication access, medication reconciliation, and rapid and ongoing primary care follow-up after hospital discharge. The intervention will be provided for one-year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Med AAAction intervention (Active Comparator): The Med AAAction intervention will include the following components: 1) medications with zero copay, 2) bedside delivery and subsequent home delivery of medications, and 3) care coordination provided by certified pharmacy technicians/health coaches to assist with medication access, medication reconciliation, and rapid and ongoing primary care follow-up after hospital discharge. The intervention will be provided for one-year.
  Interventions: Other: Med AAAction intervention
- Usual care Intervention (Placebo Comparator): As part of the usual care, the participating hospitals provide medication reconciliation services before hospital discharge. Usual care may also include MTM services for patients discharged on specialty medications or Medicare beneficiaries. Patients in both groups will receive financial incentives for completing their baseline survey ($15), and 3-month ($15), 6-month ($15), and 12-month ($25) follow-up visits.
  Interventions: Other: Med AAAction intervention

INTERVENTIONS:
Other: Med AAAction intervention — The Med AAAction intervention will include the following components: 1) medications with zero copay, 2) bedside delivery and subsequent home delivery of medications, and 3) care coordination provided by certified pharmacy technicians/health coaches to assist with medication access, medication reconciliation, and rapid and ongoing primary care follow-up after hospital discharge. The intervention will be provided for one-year.

SUMMARY:
Socioeconomically disadvantaged populations with multiple chronic conditions have high rates of nonadherence to essential chronic disease medications after hospital discharge. Medication nonadherence after hospital discharge is significantly associated with increased mortality and higher rates of readmissions and costs among these patients. Major patient-reported barriers to essential medication use after hospital discharge among low-income individuals are related to social determinants of health (SDOH) and include: 1) financial barriers , 2) transportation barriers, and 3) system-level barriers. Although, medication therapy management services are important during care transitions, these services have not proven effective in improving medication adherence after hospital discharge, highlighting a critical need for innovative interventions. The Medication Affordability, Accessibility, and Availability in Care Transitions (Med AAAction) Study will test the effectiveness of a pharmacy-led care transitions intervention versus usual care through a pragmatic randomized controlled trial of 388 Medicaid and uninsured hospital in-patients with MCC from three large healthcare systems in Tennessee. The intervention will involve: 1) medications with zero copay, 2) bedside delivery then home delivery of medications, and 3) care coordination provided by certified pharmacy technicians/health coaches to assist with medication access, medication reconciliation, and rapid and ongoing primary care follow-up. We will examine the impact of the intervention during 12 months on 1) medication adherence (primary outcome) and 2) rapid primary care follow-up, 30-day readmissions, hospitalizations and emergency department visits, and costs. We will conduct key informant interviews to understand patient experience with the acre received during and after care transitions. By examining effectiveness of the intervention on outcomes including medication adherence, health care utilization, costs, and patient experience, this study will provide valuable results to health systems, payers, and policymakers to assist in future implementation and sustainability of the intervention for socioeconomically disadvantaged populations.

DETAILED DESCRIPTION:
Care transitions are a critical time for managing medications. Socioeconomically disadvantaged populations with multiple chronic conditions (MCC) and polypharmacy have high rates of medication discrepancies and nonadherence to essential chronic disease medications following hospitalization. Medication nonadherence after hospital discharge is significantly associated with increases in readmissions, costs, and mortality among patients with MCC. Barriers to medication adherence for low-income patients are particularly acute during care transitions from the hospital to the community setting, where patients experience difficulties accessing and affording essential medications. Studies including our own, have shown that major patient-reported barriers to essential medication use after hospital discharge among low-income, primarily African American individuals are related to social determinants of health (SDOH) and include: 1) financial barriers (i.e., inability to afford medications), 2) transportation barriers (i.e., inability to access prescribed medications or needed follow-up care), and 3) system-level barriers (i.e., lack of availability of discharge medications and care coordination services to ensure rapid primary care follow-up).

Although medication therapy management (MTM) and medication reconciliation services are important during care transitions, these services have not proven effective in improving essential medication use and adherence after hospital discharge, highlighting a critical need for innovative interventions that address the major barriers to adherence following hospitalization. The PI Dr. Surbhi's pilot research has demonstrated the feasibility and potential to improve medication adherence among adult Medicaid and uninsured inpatients by directly addressing these barriers through full medication subsidy and bedside and subsequent home delivery of medications. Additionally, our previous research demonstrates that care coordination services provided by pharmacy technicians trained as coaches effectively increases rapid primary care follow-up after hospital discharge and has potential to help improve medication adherence. However, the effectiveness of interventions that directly address affordability, accessibility, and availability to improve post-discharge medication adherence in vulnerable populations is still unknown.

The Medication Affordability, Accessibility, and Availability in Care Transitions (Med AAAction) Study will examine the effectiveness of a pharmacy-led care transitions intervention versus usual care through a pragmatic randomized controlled trial of 388 Medicaid and uninsured hospital inpatients with MCC from three large non-profit healthcare systems serving a disproportionate share of low-income patients in Tennessee. The Med AAAction intervention will consist of the following components: 1) medications with zero copay, 2) bedside delivery and subsequent home delivery of medications, and 3) care coordination provided by certified pharmacy technicians/health coaches to assist with medication access, medication reconciliation, and rapid and ongoing primary care follow-up after hospital discharge. Furthermore, to understand patient experience with the care received during and after care transitions, we will obtain qualitative data through interviews with patients enrolled in the study. This study has a long-term goal to demonstrate the effectiveness of a care transitions adherence intervention model for vulnerable populations that can be readily adopted and sustained by health care delivery systems across the US. The specific aims are as follows:

Aim 1: To test the effectiveness of the intervention on essential chronic disease medication adherence (primary outcome) assessed by pill counts and a patient-reported adherence scale. Hypothesis: Intervention group participants will have higher mean adherence at 12 months compared with those randomized to the usual care.

Aim 2: To test the effectiveness of the intervention on following secondary outcomes:

Aim 2a. Health care utilization outcomes including: 1) primary care follow-up within 14 days of hospital discharge, 2) 30-day readmissions, 3) overall and preventable hospitalizations at one year, and 4) overall and preventable emergency department (ED) visits at one year using Tennessee Medicaid claims data and electronic medical records. Hypothesis: Intervention group participants will be more likely to have rapid primary care follow-up, less likely to have 30-day readmissions, and will have lower incidence of hospitalizations and ED visits over a one-year period compared with those randomized to usual care.

Aim 2b: Net cost savings associated with avoidable hospitalization and ED visits. Hypothesis: The intervention group will incur lower costs compared to usual care.

Aim 3: To understand study participants' experience with the intervention received during and after care transitions using qualitative key informant interviews.

Impact: By examining the effects of the intervention on medication adherence, health care utilization, costs, and patient experience, the study will provide valuable results to help health systems, payers, and policymakers achieve the Triple Aim - improving health outcomes and patient experience and reducing costs, among socioeconomically disadvantaged populations.

ELIGIBILITY:
Inclusion Criteria:

* Medicaid or uninsured inpatients
* 21 years or older
* ≥2 of the complex chronic conditions during index admission or prescribed/using ≥2 chronic medications for these conditions
* Patients receiving chronic disease medications from the hospital pharmacy.
* Patients will be eligible if they have multiple complex chronic conditions including diabetes, hypertension, high cholesterol, coronary artery disease, congestive heart failure, chronic lung disease, chronic kidney disease, arrhythmia, stroke, psychiatric disorders including depression and anxiety, or who are prescribed or using anticoagulants.

Exclusion Criteria:

* Medicare and Medicaid dual eligible patients.
* If the primary reason for the index admission is related to cancer, pregnancy, or a surgical procedure for an acute problem
* If patients have diagnoses of active psychosis, substance abuse, or suicidal ideation during the index admission.
* If the planned discharge location is not home.
* If patients are part of an existing pharmacy discharge program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2024-04-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Adherence to chronic disease medications | Adherence measured at 3, 6, 9, and 12 months
  Adherence to oral chronic disease medications will be assessed for the groups every 3 months using the pill count method (primary method). Additionally, we will measure patient self-reported adherence to chronic disease medications at 3-month, 6-month, and 12-month follow-up by using the following question "On how many of the last seven days, did you take your recommended medication" for each of their chronic disease medications (secondary method).

SECONDARY OUTCOMES:
Health care utilization | 12 months
  Short-term utilization outcomes will include primary care follow-up within 14 days of hospital discharge and 30-day readmissions, measured as binary outcomes (Y/N). Long-term utilization outcomes will include number of overall and preventable hospitalizations and ED visits assessed in the 12-month follow-up period. Observation visits will be combined with inpatient visits.
Cost | 12 months
  Costs will be assessed from the health system and payer perspectives. We will estimate the incremental net costs of the Med AAAction intervention compared to the usual care at each site over the period of the study. Our calculation will include both implementation costs and costs associated with hospitalizations and ED in the 12 months follow-up period. To determine costs associated with inpatient and ED visits, we will use results from Aim 2 to calculate total number of inpatient and ED visits in 12 months. For TennCare patients, we will use payment records from the claims data to estimate cost. For uninsured patients, we will use average reimbursement rates (charges) from TennCare to calculate costs for uninsured patients.
Qualitative Evaluation | 1 month and 12 month
  We will conduct key informant interviews with participants in the intervention group at two timepoints during the study. The first timepoint will include participants who completed 1 month in the program. The second timepoint will be after the participants have completed 12 months in the program. Interviews conducted at 1 months will explore the patient experience with the intervention in the hospital and post-discharge and is designed to help assess the consistency in the delivery of the intervention and enable modifications or tailoring of the intervention, based on contextual factors, if needed. Interviews at 12 months will provide a similar assessment of the participant's experience and implementation of the intervention during the period where the participant is at home.

CONTACTS AND LOCATIONS:
Overall Officials: Satya Surbhi, PhD, Principal Investigator — UTHSC
Locations (2):
- United States (2):
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - University of Tennessee Health Science Center/Regional One Health, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No